CLINICAL TRIAL: NCT01021046
Title: Deep Anterior Lamellar Keratoplasty Using Acellular Corneal Tissue Promotes Corneal Allograft Survival in High Risk Patients
Brief Title: Deep Anterior Lamellar Keratoplasty (DALK) Using Acellular Corneal Tissue Promotes Corneal Allograft Survival in High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Wei Chen, Eye Hospital, Wenzhou Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2006-11

CONDITIONS: Glycerin Cryopreserved Acellular Corneal Tissue; Deep Anterior Lamellar Keratoplasty; High Risk Keratoplasty
Keywords: deep anterior lamellar keratoplasty; rejection; high risk patients; acellular corneal tissue
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GCCT,corneal allograft survival ,DALK (Experimental): experimental group: deep anterior lamellar keratoplasty using glycerin-cryopreserved corneal tissue
  Interventions: Procedure: DALK using GCCT
- FCT,corneal allograft survival ,DALK (Experimental): control group: deep anterior lamellar keratoplasty using fresh corneal tissue
  Interventions: Procedure: DALK using FCT

INTERVENTIONS:
Procedure: DALK using GCCT — Deep anterior lamellar keratoplasty (DALK) using glycerin-cryopreserved corneal tissue
  Other Names: acellular tissue
  Arms: GCCT,corneal allograft survival ,DALK
Procedure: DALK using FCT — Deep anterior lamellar keratoplasty (DALK) using fresh corneal tissue
  Arms: FCT,corneal allograft survival ,DALK

SUMMARY:
The purpose of this study is to study whether deep anterior lamellar keratoplasty (DALK) using acellular tissue will promote corneal graft survival in high risk patients.

ELIGIBILITY:
Inclusion Criteria:

* severe bacterial keratitis
* Herpes simplex keratitis
* severe fungal keratitis
* partial limbal deficiency after chemical burn

Exclusion Criteria:

* posterior stroma involved in severe bacterial and fungal keratitis
* dry eye
* glaucoma or intraocular pressure greater than 21 mmHg
* amblyopia
* retinal abnormalities
* patients with severe systemic diseases not good for ocular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
rejection

SECONDARY OUTCOMES:
laser scanning in vivo confocal microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, MD,PhD, Principal Investigator — Eye Hospital, Wenzhou Medical College, China
Locations (1):
- Eye Hospital, Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Li J, Yu L, Deng Z, Wang L, Sun L, Ma H, Chen W. Deep anterior lamellar keratoplasty using acellular corneal tissue for prevention of allograft rejection in high-risk corneas. Am J Ophthalmol. 2011 Nov;152(5):762-70.e3. doi: 10.1016/j.ajo.2011.05.002. Epub 2011 Jul 30. PMID 21803324